CLINICAL TRIAL: NCT05088538
Title: The Effect of Quick Response (QR) Coded Teaching Plan, Prepared According to Health Literacy Levels of Patients With Total Knee Replacement Surgery, on Recovery Process and Quality of Life
Brief Title: The Effect of Quick Response Coded Teaching Plan, Patients With Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozok University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nilgun Ozbas, Assistant Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 114/05
Record Dates: First submitted 2021-09-12; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Total Knee Replacement Surgery; Patient Education
Keywords: Total knee replacement; Patient education; QR code; Health literacy; Nursing; Quality of life
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The assignment to the groups will be carried out by an independent researcher, and the group will be notified via telephone after the practitioner researcher has approved, evaluated the criteria and performed the pre-tests. At the same time, groups will be named A and B and researchers will be blinded during statistical analysis and reporting.It will not be disclosed to the participants and their caregivers in which group they belong. Surveys will be filled in by a different independent researcher blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): When the patients are in clinic,The Patient Information Form,Turkey Health Literacy Scale-32,Patient Learning Needs Scale,Functional Assessment Form,Knee Assessment Questionnaire and Quality of Life Scale Form will be filled.The second interview will be conducted on the second or third day after the surgery, just before the patients will be discharged.The Functional Assessment Form,Knee Assessment Questionnaire,Discharge Data Collection Form, and Quality of Life Questionnaire will be applied.The third interview will be performed 15 days after the surgery when the patients come for control or by phone.The 15th Day Recovery Process Data Collection Form and Knee Assessment Questionnaire will be applied.The last interview will be carried out six weeks after the surgery,either face-to-face or by phone,and the Functional Assessment Form,Knee Assessment Questionnaire, 6th Week Post-Discharge Recovery Process Data Collection Form,and Quality of Life Questionnaire will be applied again.
- Intervention group (Experimental): Unlike the control group, the intervention group will be given the education plan prepared by the researchers.
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: Patient Education — After completing the necessary forms, it is planned to give the QR-coded education booklet prepared by the researcher to the patients and to inform the patients and their relatives about the use of QR codes. At that time, it is planned that the teaching will be carried out using various training methods such as lecture, question-answer, demonstration and practice. It is thought that the teaching will be divided into 3 parts: pre-operative, post-operative and discharge. According to the physical conditions of the clinic, it is planned to provide patient education in an suitable area for teaching as much as possible. Patients will be reminded that they can access the information whenever they want and as many times as they want by scanning the QR code from their phone.
  Arms: Intervention group

SUMMARY:
With the developments in the field of health, Total Knee Replacement (TKR) surgeries are performed by applying evidence-based rapid recovery programs in many hospitals and patients can be discharged in a very short time. This situation imposes more responsibilities on patients and their relatives, especially in the post-operative period, for undertaking care, managing developing health-related conditions, and advancing the treatment process in a positive way. For this reason, it is very important for patients and their relatives to receive training before discharge on issues such as adaptation to daily life, movement, self-care skills, and complications related to post-operative home care. The fact that patients who have TKR surgery are mostly elderly individuals also increases the importance of the subject. At the same time, in order for patient education to be effective, it is very important that the information given is suitable for the level of health literacy, easily readable and understandable in a way that patients can understand. If the transmitted information is not presented in an easy and understandable way, the musculoskeletal functions, quality of life and socio economic productivity of the patients after the surgery will be endangered. In addition, patient education given to patients is not only written; Using visual, auditory and technological materials such as various presentations, videos, photographs, in accordance with different learning styles, provides a more effective coping with the problems in the post-operative period and reduces physical and psychological problems. In this context, it is seen that the use of QR code, which is a digital technological application that has recently been used in the field of health, is an application that can provide an easier understanding of the information transmitted verbally and in writing by healthcare professionals.

DETAILED DESCRIPTION:
Individuals who have undergone TKR surgery want to receive information about many subjects such as patient education, recovery, home care, surgery, movement, pain, exercise, walking, nutrition, working life, weight control, illness, complications. It is very important that the information is appropriate for the level of health literacy and that it is provided not only by written but also by various visual, auditory and technological methods in order to effectively transfer the information needed by the patients during the challenging process that significantly affects their mobility and daily living activities. This study was planned as a randomized controlled study in order to examine the effect of the rapid response QR coded teaching plan prepared according to the health literacy levels of the patients who had TKR surgery on the healing process and quality of life.

Hypotheses of the study:

H1a- Patient education with QR code, which is planned according to health literacy levels, positively affects patients' quality of life.

H1b- Patient education with QR code, which is planned according to health literacy levels, reduces patients' problems on the 15th day after surgery.

H1c- Patient education with QR code, which is planned according to health literacy levels, reduces patients' problems in the 6th week after surgery.

H1d- Patient education with QR code, which is planned according to health literacy levels, affects the postoperative improvement in functional status in patients.

Type of Study: Randomized controlled trial

Method:

102 (51 intervention, 51 control) patients who underwent TKR surgery will be randomized and divided into two groups as intervention and control groups. No intervention will be made to the patients in the control group and the patients will receive routine treatment and care in the clinic. In addition to the routine treatment and care, the patients in the intervention group will be taught with a QR code prepared by the researcher. Data will be collected using the Patient Identification Form, The Patient Learning Needs Scale, Functional Assessment Form, Knee Assessment Questionnaire, Turkish Health Literacy Scale-32, Discharge Data Collection Form, Post-Discharge Day 15 of the Healing Process Data Collection Form, Post-Discharge Week 6 of the Healing Process Data Collection Form and the Quality of Life Scale.

While evaluating the data, it is planned to be analyzed as randomized.It is planned to use multiple completion methods when there are missing data.

Statistical analyzes are planned to be evaluated with the Statistical Package for the Social Sciences (SPSS)-24 package program. It is planned to use frequency charts and descriptive statistics in order to interpret the data, parametric techniques for normal distributions and non-parametric techniques for non-normal distributions.

ELIGIBILITY:
Inclusion Criteria:

* Not having knee replacement surgery before
* Not having a history of psychiatric problems
* Having known how to read and write
* Having a smart phone
* Having internet access on the phone
* Having been agreed to participate in the research

Exclusion Criteria:

* Having previous knee replacement surgery
* Having a history of psychiatric problems
* Not having known how to read and write
* Not having a smart phone
* Not having internet access on the phone
* Not having been agreed to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
The Quality of Life Scale Change (SF-36) | 1st day of admission to the clinic change the quality of life score at before intervention, change from baseline the quality of lıfe score at 3rd postoperative day, change from baseline the quality of life score at 6th postoperative week
  The Quality of Life Scale (SF-36), one of the most used scales to measure quality of life; It is a self-assessment scale that can be filled in a short time and is highly sensitive.While applying the scale, individuals are asked to answer considering the last 4 weeks. The scale consists of 36 questions and 8 sub-parameters (body pain, limitation due to physical problems, limitation due to mental problems, mental well-being, fatigue, general health perception, social function and physical function). In scoring, each parameter is evaluated between 0 and 100 points. A score of 0 indicates poor health, and a score of 100 indicates good health. The higher the score, the higher the quality of life.

SECONDARY OUTCOMES:
The Function Evaluation Form Change | 1st day of admission to the clinic change the function evaluation score at before intervention, change from baseline function evaluation score at 3rd postoperative day, change from baseline function evaluation score at 6th postoperative week
  The Functional Evaluation Form was developed to determine the functional status of patients who had TKR surgery and hip replacement surgery. The form consists of 8 sections and each section is scored within itself. The highest possible score is 100. The increase in score indicates the improvement in the functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Özbaş, Assist Prof, Principal Investigator — Bozok University; Ahmet Acar, Doctor, Study Chair — Dışkapı Yıldırım Beyazıt Training and Research Hospital
Locations (1):
- Dışkapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No